CLINICAL TRIAL: NCT00807885
Title: INcreased Flow Utilizing Subcutaneously-Enabled Fluids Administration Technique Study (INFUSE-AT): A Randomized, Open-Label, Parallel Group, Phase IV, Study Evaluating the Techniques of Administration of Subcutaneous Fluids Enabled by Human Recombinant Hyaluronidase (Hylenex) in Healthy Adult Volunteers
Brief Title: Study of Techniques of Subcutaneous Administration of Fluids Enabled by Human Recombinant Hyaluronidase
Acronym: INFUSE-AT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Baxter Healthcare Corporation (Industry)
Collaborators: Halozyme Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1838-007
Record Dates: First submitted 2008-12-10; First posted 2008-12-12 (Estimated); Results first posted 2011-10-18 (Estimated); Last update posted 2011-10-26 (Estimated); Status verified 2011-10

CONDITIONS: Dehydration
Keywords: dehydration; fluid therapy; hyaluronoglucosaminidase; hyaluronidase; hypodermoclysis; clysis; subcutaneous hydration; subcutaneous rehydration; hyaluronan; rHuPH20
MeSH Terms: conditions — Dehydration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (9):
- Tegaderm-secured 24 ga Teflon catheter (Experimental): subcutaneous administration of a single 150 U dose of hylenex, followed by subcutaneous infusion (delivered by large volume infusion pump) of 1000 mL Lactated Ringer's solution, both delivered through a 24-gauge, 0.75 inch long, Teflon angiocatheter secured with Tegaderm
  Interventions: Drug: hylenex-facilitated subcutaneous Lactated Ringer's infusion
- Tape-secured 24 ga Teflon catheter (Experimental): subcutaneous administration of a single 150 U dose of hylenex, followed by subcutaneous infusion (delivered by large volume infusion pump) of 1000 mL Lactated Ringer's solution, both delivered through a 24-gauge, 0.75 inch long, Teflon angiocatheter secured with a tape double chevron
  Interventions: Drug: hylenex-facilitated subcutaneous Lactated Ringer's infusion
- Tegaderm-secured 24 ga polyurethane catheter (Experimental): subcutaneous administration of a single 150 U dose of hylenex, followed by subcutaneous infusion (delivered by large volume infusion pump) of 1000 mL Lactated Ringer's solution, both delivered through a 24-gauge, 0.75 inch long, polyurethane angiocatheter secured with Tegaderm
  Interventions: Drug: hylenex-facilitated subcutaneous Lactated Ringer's infusion
- Tape-secured 24 ga polyurethane catheter (Experimental): subcutaneous administration of a single 150 U dose of hylenex, followed by subcutaneous infusion (delivered by large volume infusion pump) of 1000 mL Lactated Ringer's solution, both delivered through a 24-gauge, 0.75 inch long, polyurethane angiocatheter secured with a tape double chevron
  Interventions: Drug: hylenex-facilitated subcutaneous Lactated Ringer's infusion
- Tegaderm-secured 20 ga Teflon catheter (Experimental): subcutaneous administration of a single 150 U dose of hylenex, followed by subcutaneous infusion (delivered by large volume infusion pump) of 1000 mL Lactated Ringer's solution, both delivered through a 20-gauge, 1.0 inch long, Teflon angiocatheter secured with Tegaderm
  Interventions: Drug: hylenex-facilitated subcutaneous Lactated Ringer's infusion
- Tape-secured 20 ga Teflon catheter (Experimental): subcutaneous administration of a single 150 U dose of hylenex, followed by subcutaneous infusion (delivered by large volume infusion pump) of 1000 mL Lactated Ringer's solution, both delivered through a 20-gauge, 1.0 inch long, Teflon angiocatheter secured with a tape double chevron
  Interventions: Drug: hylenex-facilitated subcutaneous Lactated Ringer's infusion
- Tegaderm-secured 20 ga polyurethane catheter (Experimental): subcutaneous administration of a single 150 U dose of hylenex, followed by subcutaneous infusion (delivered by large volume infusion pump) of 1000 mL Lactated Ringer's solution, both delivered through a 20-gauge, 1.0 inch long, polyurethane angiocatheter secured with Tegaderm
  Interventions: Drug: hylenex-facilitated subcutaneous Lactated Ringer's infusion
- Tape-secured 20 ga polyurethane catheter (Experimental): subcutaneous administration of a single 150 U dose of hylenex, followed by subcutaneous infusion (delivered by large volume infusion pump) of 1000 mL Lactated Ringer's solution, both delivered through a 20-gauge, 1.0 inch long, polyurethane angiocatheter secured with a tape double chevron
  Interventions: Drug: hylenex-facilitated subcutaneous Lactated Ringer's infusion
- SC button with 27 ga X 9 mm needle (Experimental): subcutaneous administration of a single 150 U dose of hylenex, followed by subcutaneous infusion (delivered by large volume infusion pump) of 1000 mL Lactated Ringer's solution, both delivered through a button-type subcutaneous delivery system (with a 27-gauge, 9 mm long metal needle)
  Interventions: Drug: hylenex-facilitated subcutaneous Lactated Ringer's infusion

INTERVENTIONS:
Drug: hylenex-facilitated subcutaneous Lactated Ringer's infusion — single subcutaneous 150 U dose of hylenex, followed by subcutaneous infusion of 1000 mL Lactated Ringer's solution
  Other Names: hylenex; rHuPH20; LR; LR solution

SUMMARY:
The purpose is to evaluate the ease of use and technical challenges encountered during subcutaneous infusion of Lactated Ringer's (LR) solution, preceded by recombinant human hyaluronidase (hylenex), utilizing commonly used angiocatheter gauges and button delivery systems. The safety and tolerability of hylenex-augmented SC infusion of LR through these delivery systems is also being evaluated.

ELIGIBILITY:
Inclusion Criteria:

* male or female, aged 18 to 60 years
* intact normal skin without potentially obscuring features on both anterior thighs in the area intended for infusion
* agreeing to no fluid intake for 12 hours prior to start of study infusion
* vital signs within normal range or, if outside normal range, deemed not clinically significant
* metabolic panel, hematology, virology and standard 10-test urine dipstick tests within normal range, or if outside normal range, deemed not clinically significant
* if female of child-bearing potential,negative serum pregnancy tests
* negative urine drug screens
* written informed consent for participation

Exclusion Criteria:

* lower extremity edema
* lower extremity pathology that could interfere with study outcome
* history of cardiovascular disease
* rales on lung auscultation
* known allergy to hyaluronidase or other ingredient in the formulation of hylenex
* pregnancy or breast-feeding a child
* exposure to any experimental drug within 30 days prior to study participation
* previous participation in this study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2008-12; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George Harb, MD, MPH, Study Director — Baxter Healthcare Corporation
Locations (2):
- United States (2):
  - MDS Pharma Services, Lincoln, Nebraska
  - MDS Pharma Services, Neptune City, New Jersey

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tegaderm-secured 24 ga Teflon Catheter | Tape-secured 24 ga Teflon Catheter | Tegaderm-secured 24 ga Polyurethane Catheter | Tape-secured 24 ga Polyurethane Catheter | Tegaderm-secured 20 ga Teflon Catheter | Tape-secured 20 ga Teflon Catheter | Tegaderm-secured 20 ga Polyurethane Catheter | Tape-secured 20 ga Polyurethane Catheter | SC Button With 27 ga X 9 mm Needle
Started | 10 | 11 | 11 | 10 | 12 | 12 | 12 | 11 | 11
Completed | 10 | 11 | 11 | 10 | 12 | 11 (Subject completed treatment, but lost to follow-up) | 12 | 11 | 11
Not Completed | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tegaderm-secured 24 ga Teflon Catheter | Tape-secured 24 ga Teflon Catheter | Tegaderm-secured 24 ga Polyurethane Catheter | Tape-secured 24 ga Polyurethane Catheter | Tegaderm-secured 20 ga Teflon Catheter | Tape-secured 20 ga Teflon Catheter | Tegaderm-secured 20 ga Polyurethane Catheter | Tape-secured 20 ga Polyurethane Catheter | SC Button With 27 ga X 9 mm Needle | Total
Number analyzed (Participants) | 10 | 11 | 11 | 10 | 12 | 12 | 12 | 11 | 11 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 11 | 11 | 10 | 12 | 12 | 12 | 11 | 11 | 100
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 34.6 (9.39) | 36.0 (10.6) | 33.8 (10.4) | 35.3 (10.9) | 34.0 (12.5) | 34.3 (10.3) | 33.6 (10.7) | 32.4 (12.7) | 36.6 (12.3) | 34.5 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 8 | 3 | 3 | 6 | 5 | 4 | 5 | 38
  Male | 7 | 10 | 3 | 7 | 9 | 6 | 7 | 7 | 6 | 62
Region of Enrollment [Number; unit: participants]
  United States | 10 | 11 | 11 | 10 | 12 | 12 | 12 | 11 | 11 | 100

OUTCOME MEASURES:

1. Primary Outcome: Technical Challenges
Description: Protocol-specified challenges encountered during subcutaneous (SC) hylenex administration and/or SC infusion of Lactated Ringer's solution, including SC catheter kinking, catheter/button dislodgement, catheter/button pull-out, infusion pump alarm, other pump failure, healthcare provider intervention to secure/maintain SC infusion eg, re-taping, catheter/button manipulation, etc, and any other type of technical challenge encountered
Time Frame: throughout subcutaneous hylenex and fluid administration period (continuous)
Population: ITT (all treated subjects)
Measure: Number; unit: participants
Arm/Group | Tegaderm-secured 24 ga Teflon Catheter | Tape-secured 24 ga Teflon Catheter | Tegaderm-secured 24 ga Polyurethane Catheter | Tape-secured 24 ga Polyurethane Catheter | Tegaderm-secured 20 ga Teflon Catheter | Tape-secured 20 ga Teflon Catheter | Tegaderm-secured 20 ga Polyurethane Catheter | Tape-secured 20 ga Polyurethane Catheter | SC Button With 27 ga X 9 mm Needle
Number analyzed (Participants) | 10 | 11 | 11 | 10 | 12 | 12 | 12 | 11 | 11
participants
  Subjects with at Least One Technical Challenge | 2 | 3 | 2 | 2 | 2 | 2 | 3 | 2 | 3
  Subjects with No Technical Challenges | 8 | 8 | 9 | 8 | 10 | 10 | 9 | 9 | 8
  Subjects with 1 TEchnical Challenge | 2 | 3 | 2 | 1 | 2 | 2 | 3 | 0 | 3
  Subjects with 2 Technical Challenges | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
  Subjects with 3 Technical Challenges | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Subjects with Catheter Kinking | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 2 | 0
  Subjects with Catheter Dislodgement | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Subjects with Catheter Pulled Out | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Subjects with Infusion Pump Alarm | 2 | 2 | 2 | 1 | 2 | 2 | 3 | 1 | 3
  Subjects with Infusion Pump Failure | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Attempts Needed to Successfully Place Subcutaneous Catheter/Button
Time Frame: from start of first attempt until completion of catheter/button placement
Population: ITT (all treated subjects)
Measure: Number; unit: participants
Arm/Group | Tegaderm-secured 24 ga Teflon Catheter | Tape-secured 24 ga Teflon Catheter | Tegaderm-secured 24 ga Polyurethane Catheter | Tape-secured 24 ga Polyurethane Catheter | Tegaderm-secured 20 ga Teflon Catheter | Tape-secured 20 ga Teflon Catheter | Tegaderm-secured 20 ga Polyurethane Catheter | Tape-secured 20 ga Polyurethane Catheter | SC Button With 27 ga X 9 mm Needle
Number analyzed (Participants) | 10 | 11 | 11 | 10 | 12 | 12 | 12 | 11 | 11
participants
  1 Attempt | 10 | 11 | 10 | 10 | 12 | 11 | 12 | 11 | 11
  2 Attempts | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0

3. Secondary Outcome: Time Needed to Successfully Place Subcutaneous Catheter/Button
Time Frame: from start of first attempt until completion of catheter/button placement
Population: ITT (all treated subjects)
Measure: Median (Full Range); unit: seconds
Arm/Group | Tegaderm-secured 24 ga Teflon Catheter | Tape-secured 24 ga Teflon Catheter | Tegaderm-secured 24 ga Polyurethane Catheter | Tape-secured 24 ga Polyurethane Catheter | Tegaderm-secured 20 ga Teflon Catheter | Tape-secured 20 ga Teflon Catheter | Tegaderm-secured 20 ga Polyurethane Catheter | Tape-secured 20 ga Polyurethane Catheter | SC Button With 27 ga X 9 mm Needle
Number analyzed (Participants) | 10 | 11 | 11 | 10 | 12 | 12 | 12 | 11 | 11
seconds | 23 [1 to 39] | 43 [2 to 84] | 30 [2 to 63] | 34 [10 to 96] | 30 [2 to 58] | 49 [2 to 133] | 31 [1 to 90] | 15 [1 to 96] | 9 [1 to 47]

4. Secondary Outcome: Time Required to Infuse 1000 mL Fluid
Time Frame: from start of Lactated Ringer's (LR) infusion until 1000 mL LR infused
Population: ITT (all treated subjects)
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Tegaderm-secured 24 ga Teflon Catheter | Tape-secured 24 ga Teflon Catheter | Tegaderm-secured 24 ga Polyurethane Catheter | Tape-secured 24 ga Polyurethane Catheter | Tegaderm-secured 20 ga Teflon Catheter | Tape-secured 20 ga Teflon Catheter | Tegaderm-secured 20 ga Polyurethane Catheter | Tape-secured 20 ga Polyurethane Catheter | SC Button With 27 ga X 9 mm Needle
Number analyzed (Participants) | 10 | 11 | 11 | 10 | 12 | 12 | 12 | 11 | 11
hours | 6.82 (0.058) | 6.78 (0.098) | 6.81 (0.013) | 6.80 (0.114) | 6.78 (0.071) | 6.80 (0.013) | 6.81 (0.078) | 6.79 (0.108) | 6.82 (0.078)

ADVERSE EVENTS:
Time Frame: 6 d post-treatment
Arm/Group | Tegaderm-secured 24 ga Teflon Catheter | Tape-secured 24 ga Teflon Catheter | Tegaderm-secured 24 ga Polyurethane Catheter | Tape-secured 24 ga Polyurethane Catheter | Tegaderm-secured 20 ga Teflon Catheter | Tape-secured 20 ga Teflon Catheter | Tegaderm-secured 20 ga Polyurethane Catheter | Tape-secured 20 ga Polyurethane Catheter | SC Button With 27 ga X 9 mm Needle
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/11 | 0/11 | 0/10 | 1/12 | 0/12 | 0/12 | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 6/10 | 5/11 | 9/11 | 7/10 | 9/12 | 10/12 | 10/12 | 10/11 | 8/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tegaderm-secured 24 ga Teflon Catheter (N=10) | Tape-secured 24 ga Teflon Catheter (N=11) | Tegaderm-secured 24 ga Polyurethane Catheter (N=11) | Tape-secured 24 ga Polyurethane Catheter (N=10) | Tegaderm-secured 20 ga Teflon Catheter (N=12) | Tape-secured 20 ga Teflon Catheter (N=12) | Tegaderm-secured 20 ga Polyurethane Catheter (N=12) | Tape-secured 20 ga Polyurethane Catheter (N=11) | SC Button With 27 ga X 9 mm Needle (N=11)
calculus ureteric (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 — Unrelated to treatment
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tegaderm-secured 24 ga Teflon Catheter (N=10) | Tape-secured 24 ga Teflon Catheter (N=11) | Tegaderm-secured 24 ga Polyurethane Catheter (N=11) | Tape-secured 24 ga Polyurethane Catheter (N=10) | Tegaderm-secured 20 ga Teflon Catheter (N=12) | Tape-secured 20 ga Teflon Catheter (N=12) | Tegaderm-secured 20 ga Polyurethane Catheter (N=12) | Tape-secured 20 ga Polyurethane Catheter (N=11) | SC Button With 27 ga X 9 mm Needle (N=11)
Infusion site erythema (General disorders) | 3 | 2 | 4 | 2 | 2 | 3 | 2 | 4 | 3
Infusion site pain (General disorders) | 2 | 4 | 4 | 3 | 6 | 9 | 8 | 8 | 3
Infusion site swelling (General disorders) | 0 | 1 | 1 | 2 | 3 | 4 | 3 | 0 | 1
Headache (Nervous system disorders) | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 3 | 1 | 2 | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
For this study, Baxter requires a review of any planned PI results communications (eg, for confidential information) up to 90 days prior to submission or communication. Baxter may request an additional delay of up to 60 days (eg, to allow for intellectual property protection).